CLINICAL TRIAL: NCT06150300
Title: STAPLE (Severe asThmA PuLmonary rEhab): Examining the Effects of a Remote Pulmonary Rehabilitation Program in the Severe Asthma Population.
Brief Title: Examining the Effects of a Remote Pulmonary Rehabilitation Program in the Severe Asthma Population.
Acronym: STAPLE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Brianne Philipenko, Assistant Professor, MD FRCPC, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bio4357
Record Dates: First submitted 2023-11-20; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity intervention (Active Comparator): 8 week virtual pulmonary rehab program including breathing exercises and educational messages.
  Interventions: Behavioral: Pulmonary rehab program
- Placebo (Placebo Comparator): Breathing exercises and educational messages
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Pulmonary rehab program — Exercise videos, breathing exercises, and educational messages delivered virtually
  Arms: Physical activity intervention
Behavioral: Placebo — Breathing exercises and educational messages
  Arms: Placebo

SUMMARY:
This is a randomized control trial evaluating the effect of a novel mobile application-delivered pulmonary rehabilitation program in adult severe asthma patients. The intervention will include eight weeks of exercise videos that progress in difficulty, as well as asthma-specific educational content. The primary outcome measure is change in functional exercise capacity as measured by six-minute walk distance. Secondary outcome measures will include evaluation of overall feasibility, and change in CPET parameters such as VO2max. Change in asthma control questionnaire (ACQ), asthma quality of life questionnaire (AQLQ) and PRAISE self-efficacy score will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older with a diagnosis of asthma by a respirologist. They must have severe disease defined by GINA severity classification. Participants must have access to a smartphone or internet browser to allow access to study content.

Exclusion Criteria:

* Exclusion criteria include comorbid cardiopulmonary or musculoskeletal conditions that may impact exercise tolerance in accordance with the American Thoracic Society CPET guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
CPET | After 8 weeks of intervention
  VO2max

IPD SHARING:
Plan to Share IPD: No